CLINICAL TRIAL: NCT02517099
Title: Use of Pathological Phenotype to Determine Optimal Management for Moderate to Severe Preschool Wheeze
Brief Title: Preschool Wheeze: Inflammation/Infection Guided Management
Acronym: PrIGMa
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Imperial College London (Other)
Collaborators: National Institute for Health Research, United Kingdom (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 165460
Record Dates: First submitted 2015-08-04; First posted 2015-08-06 (Estimated); Results first posted 2023-03-06 (Actual); Last update posted 2023-03-06 (Actual); Status verified 2022-05

CONDITIONS: Asthma
Keywords: Preschool; Wheeze; Moderate; Severe
MeSH Terms: conditions — Asthma; Respiratory Sounds; Lymphoma, Follicular | interventions — Beclomethasone; Amoxicillin-Potassium Clavulanate Combination; Azithromycin

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- Pathological phenotype (Active Comparator): Regular inhaled steroids- Beclometasone dipropionate 200mcg bd for 4 months OR antibiotic therapy- Co- amoxiclav (0.3ml/kg bd) or Azithromycin (10mg/kg od) for 4 weeks
  Interventions: Drug: Beclometasone; Drug: Co-amoxiclav; Drug: Azithromycin
- Clinical guidelines (Active Comparator): The children will be treated as directed by their Consultant Paediatrician. The treatment may include- regular inhaled steroids- beclometasone dipropionate 200mcg bd for 4 months OR antibiotic therapy- Co-amoxiclav (0.3ml/kg bd) or Azithromycin (10mg/kg od) for 4 weeks
  Interventions: Drug: Beclometasone; Drug: Co-amoxiclav; Drug: Azithromycin

INTERVENTIONS:
Drug: Beclometasone — Beclometasone dipropionate 200mcg bd for 4 months
  Other Names: Clenil
Drug: Co-amoxiclav — Co-amoxiclav 0.3ml/kg bd for 4 weeks
  Other Names: Augmentin Duo
Drug: Azithromycin — Azithromycin 10mg/kg od for 4 weeks
  Other Names: Zithromax

SUMMARY:
This is a single-centre, randomised-controlled trial, comparing management of preschool wheeze. It specifically aims to compare management of preschool wheeze using current clinical guidelines to management determined by eosinophilic inflammation and infection. Participants will be children aged 1-5 years who have recurrent wheezing and will be allocated to one of two treatment groups, either current clinical care or pathological phenotype based management. They will be asked to make 2 study visits to the Royal Brompton Hospital over the course of 4 months.

DETAILED DESCRIPTION:
This study will determine the efficacy of treating preschool wheeze based on objective biomarkers of inflammation and presence of bacterial infection, and compare this to current clinical guidelines based management. Subjects will be recruited from out-patient clinics and attend for a screening/research visit during which assessments of pathological phenotype (bacterial infection and inflammation) will be made from induced sputum and blood. Their clinical phenotype will be determined by the Consultant. Subsequently, patients will be randomised to one of two arms:

i) current clinical care ( as directed by their Consultant) ii) pathological phenotype based management- presence of eosinophilia in blood (_> 2%) or induced sputum (>2.4%) - will receive twice daily inhaled steroids ( beclometasone 200mcg bd) for 4 months, presence of bacterial infection in induced sputum or oropharyngeal swab- will receive 4 weeks of antibiotics targeted to the isolate, IF BOTH eosinophilic inflammation AND infection are present, then inflammation alone will be treated for 4 months.

All patients will continue on as required bronchodilator therapy, and any other anti-inflammatory therapy ( other than inhaled steroids) e.g. montelukast.

All participants will undergo an initial research/screening visit which will involve the following tests:

Full blood count Total serum immunoglobulin E and radioallergosorbent test to house dust mite, grass pollen, tree pollen, cat, dog, aspergillus, milk, egg, peanut Assessment of lung function by incentive spirometry and lung clearance index (LCI) using the multiple breath washout technique Exhaled nitric oxide- using the offline tidal breathing technique Sputum induction using nebulised hypertonic saline Oro- pharyngeal swab Symptom questionnaire Health related quality of life questionnaire

Management in the pathological phenotype arm:

1. Eosinophilic inflammation, no bacterial infection:

   Children with sputum eosinophils >2.4% or blood eosinophils equal to and above 2% will be defined as eosinophilic and management will be as follows:

   i) Regular inhaled steroids ( beclometasone 200mcg bd) for 4 months in those previously not on any regular therapy.

   ii) Of children who have already been prescribed inhaled steroid therapy, those with an eosinophilic phenotype will continue for a further 4 months.

   iii) Children who have already been prescribed a regular leukotriene receptor antagonist will continue this and regular inhaled steroids (beclometasone 200mcg bd) will be added to their maintenance therapy for 4 months.

   iv) Use of as required bronchodilator therapy will continue
2. Non- eosinophilic, no inflammation, no infection:

   Children with either sputum eosinophils _<2.4% or blood eosinophils <2% will be defined as non- eosinophilic and management will be as follows:

   i) Use of as required bronchodilators for acute symptoms ii) Non- eosinophilic children that have already been prescribed regular inhaled steroids will be asked to stop them for 4 months Children with no bacterial growth from oropharyngeal swab or induced sputum, and without eosinophilic inflammation will continue management according to the non-eosinophilic, no inflammation, no infection profile.
3. Bacterial infection, no eosinophilic inflammation:

   Children with a positive bacterial culture result from oropharyngeal swab or induced sputum will be treated with a 4 week course of antibiotics. Four weeks of antibiotic therapy will be used as this has been shown to be beneficial in a previous study of severe preschool wheeze. If these children have already been prescribed regular inhaled steroids, they will be stopped for 4 months.
4. Eosinophilic inflammation AND bacterial infection:

Children with raised eosinophils in induced sputum or blood AND positive bacterial culture will be managed according to the eosinophilic inflammation alone guideline. They will only be given inhaled steroids for 4 months, and no antibiotics. This is to assess only one intervention at a time. However, the investigators do not anticipate many children will be in this group as our previous data shows those with positive bacterial cultures are very unlikely to have eosinophilia.

Management in the clinical guidelines arm:

The children will be treated as directed by their Consultant Paediatrician. The prescription for the drugs to be used will be dispensed from the pharmacy department at the Royal Brompton Hospital- as directed by the clinician. Usually only 2 weeks of medication is prescribed by the pharmacy, but for this trial 4 months' supply will be given.

Concomitant treatment

The following medication will be allowed to continue during the intervention period in both study arms:

1. Use of rescue medication with bronchodilators for acute symptoms- salbutamol and/or ipratropium bromide
2. Use of leukotriene receptor antagonist- montelukast- can continue regardless of whether it is being taken regularly or as required for acute symptoms

Monitoring:

The trial will be monitored according to the monitoring plan agreed and written by the Sponsor, based on internal risk assessment procedure. Where appropriate the CI will be asked to complete a copy of the Sponsor's self-monitoring template. It is the responsibility of the CI to ensure this is completed and submitted to the research organisation on request. It is the responsibility of the research organisation to determine the monitoring risk assessment and explain the rationale.

The study may be subject to inspection and audit by Imperial College London under their remit as Sponsor, the Study Coordination Centre and other regulatory bodies to ensure adherence to good clinical practice.

Statistics and Data analysis:

Categorical data will be presented as number and percentage and comparisons between groups done using the chi squared or Fishers exact test. All numerical data will be tested for normality and normally distributed data will be presented as mean standard deviation and comparisons between groups done using the 2 sample independent t test. For the data that are not normally distributed the median (IQR) will be presented and comparisons between groups done using the Mann-Whitney test. Poisson regression will be done to determine the factors that affect the primary endpoint, the number of unplanned hospital visits.

There will be data checks to compare data entered into the registry, against predefined rules for range using the INFORM database.

Type of subjects to be recruited:

All subjects will be aged between 1 and 5 years old. All subjects will have moderate to severe preschool wheeze, defined as _>2 oral steroid bursts for acute wheeze in the last 12 months, with at least one oral steroid burst in the last 6 months.

Number of subjects:

Based on published data for children with moderate preschool wheeze it is apparent that approximately five healthcare attendances occur per child per year. In the current study, the investigators wish to reduce the proportion of healthcare contacts by at least one-third per year. In order to achieve this with 80% power, and accepting statistical significance at the 5% level, the investigators require a minimum of 36 evaluable patients with moderate wheeze per group. Evaluable patients are those from whom at least a blood sample to assess inflammation and an oropharyngeal swab to determine infection can be obtained prior to randomisation. A total of at least 72 children will therefore be recruited. However, this is the minimum number, and the investigators aim to recruit 100 children (50 per group) if possible.

The number of subjects is not based on a precise power calculation as this is a proof of concept study to determine the feasibility of this approach, and to inform a future power calculation for a large multi-centre trial addressing the same question.

ELIGIBILITY:
Inclusion Criteria:

* Reported recurrent wheeze, needing at least 2 courses of oral steroids in the last 12 months, at least one course of oral steroids in the last 6 months
* Past wheeze confirmed by a clinician

Exclusion Criteria:

* Any known cardiac disease
* Any chronic respiratory condition (other than preschool wheeze) diagnosed by a physician
* Any chronic condition that increases susceptibility to respiratory tract infections such as severe developmental delay and feeding difficulty/unsafe swallow Prematurity <34 weeks, or requirement of ventilation in the newborn period History of neonatal chronic lung disease Family not contactable by telephone

Ages: 1 Year to 5 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 60 (Actual)
Dates: Start 2015-06-05 (Actual); Primary Completion 2018-08-17 (Actual); Study Completion 2018-08-17 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Sejal Saglani, Principal Investigator — Imperial College London
Locations (1):
- Royal Brompton Hospital, London, United Kingdom

REFERENCES:
- [Derived] Undela K, Goldsmith L, Kew KM, Ferrara G. Macrolides versus placebo for chronic asthma. Cochrane Database Syst Rev. 2021 Nov 22;11(11):CD002997. doi: 10.1002/14651858.CD002997.pub5. PMID 34807989

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Pathological Phenotype | Clinical Guidelines
Started | 30 | 30
Completed | 25 | 27
Not Completed | 5 | 3

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Pathological Phenotype | Clinical Guidelines | Total
Number analyzed (Participants) | 30 | 30 | 60
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 30 | 30 | 60
  Between 18 and 65 years | 0 | 0 | 0
  >=65 years | 0 | 0 | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 9 | 9 | 18
  Male | 21 | 21 | 42
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0
  Not Hispanic or Latino | 29 | 25 | 54
  Unknown or Not Reported | 1 | 5 | 6
Region of Enrollment [Number; unit: participants]
  United Kingdom | 30 | 30 | 60

OUTCOME MEASURES:

1. Primary Outcome: Number of Unscheduled Healthcare Visits (UHCV)
Description: Actual number of unscheduled healthcare visits (UHCV) includes GP, A&E or hospital admission. This is median number of visits in 4 months - with range.
Time Frame: 4 months
Population: 8 patients failed to attend follow up at 4 months
Measure: Median (Full Range); unit: number of visits
Arm/Group | Pathological Phenotype | Clinical Guidelines
Number analyzed (Participants) | 25 | 27
number of visits | 0.5 [0 to 7] | 0.5 [0 to 11]
Statistical Analysis 1: Comparison: Pathological Phenotype vs Clinical Guidelines; Test type: Superiority; p = 0.05, Wilcoxon (Mann-Whitney); Median Difference (Final Values) = 2.0, 95% CI 2-sided [1.591 to 8.80], Standard Error of Mean 0.384

2. Secondary Outcome: Health Related Quality of Life
Description: Quality of life assessed using the Paediatric Caregivers Asthma Quality of Life Questionnaire (PACQLQ). The scores are from 1.0-7.0, higher value is a better outcome. We calculated the actual score at baseline and at 4 months. A change in score of 0.5 is considered clinically significant. We recorded actual value at baseline and actual value at 4 months.
Time Frame: 4 months
Population: 8 patients failed to attend for 4 month follow up
Measure: Median (Full Range); unit: score on a scale
Arm/Group | Pathological Phenotype | Clinical Guidelines
Number analyzed (Participants) | 25 | 27
score on a scale | 6.7 [1.5 to 7.0] | 6.4 [2.4 to 7.0]

3. Secondary Outcome: Symptom Days
Description: Number of days with symptoms during 4 months
Time Frame: 4 months
Population: 8 patients failed to attend for 4 month follow up
Measure: Median (Full Range); unit: days
Arm/Group | Pathological Phenotype | Clinical Guidelines
Number analyzed (Participants) | 25 | 27
days | 9 [0 to 45] | 12 [0 to 49]

4. Secondary Outcome: Number of Courses of Oral Steroids
Description: Number of steroid courses needed during 4 months for any acute symptoms.
Time Frame: 4 months and up to 1 year later
Population: 8 patients failed to attend for 4 month follow up
Measure: Number; unit: number of steroid courses
Arm/Group | Pathological Phenotype | Clinical Guidelines
Number analyzed (Participants) | 25 | 27
number of steroid courses | 13 | 14

ADVERSE EVENTS:
Time Frame: Adverse event data were collected during the 4 months of the intervention period.
Description: Adverse event data were collected prospectively No significant adverse events occurred
Arm/Group | Pathological Phenotype | Clinical Guidelines
All-Cause Mortality (participants affected / at risk) | 0/30 | 0/30
Serious Adverse Events (participants affected / at risk) | 0/30 | 0/30
Other Adverse Events (participants affected / at risk) | 0/30 | 0/30

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2016-08-30): https://cdn.clinicaltrials.gov/large-docs/99/NCT02517099/Prot_SAP_000.pdf